CLINICAL TRIAL: NCT07279220
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial to Evaluate the Safety and Effectiveness of the Vascular Closure Device for Femoral Artery Hemostasis in Patients of Femoral Artery Puncture
Brief Title: Safety and Effectiveness of the Vascular Closure Device for Femoral Artery Hemostasis in Patients of Femoral Artery Puncture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Bomaian Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMA-202501
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Femoral Artery Puncture; Vascular Closure Device; Hemostasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Device: Vascular Closure Device Manufactured by Shanghai Bomaian Medical Technology Co., Ltd.
- Control Group (Active Comparator)
  Interventions: Device: MynxGrip Vascular Closure Device Manufactured by Cordis US Corp

INTERVENTIONS:
Device: Vascular Closure Device Manufactured by Shanghai Bomaian Medical Technology Co., Ltd. — The test group will use the Vascular Closure Device manufactured by Shanghai Bomaian Medical Technology Co., Ltd. for femoral artery hemostasis in patients of femoral artery puncture
  Arms: Test Group
Device: MynxGrip Vascular Closure Device Manufactured by Cordis US Corp — The control group will use MynxGrip Vascular Closure Device Manufactured by Cordis US Corp for femoral artery hemostasis in patients of femoral artery puncture
  Arms: Control Group

SUMMARY:
The purpose of this study is to verify the safety and effectiveness of the Vascular Closure Device manufactured by Shanghai Bomaian Medical Technology Co., Ltd. for femoral artery hemostasis in patients of femoral artery puncture.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~80, male or non-pregnant female;
2. Subjects undergoing interventional diagnostic or therapeutic procedures via femoral artery puncture;
3. Subjects using 5F to 8F sheaths during the procedure (Note: Subjects using 5F-7F sheaths will enter the main randomized controlled cohort, while subjects using 8F sheaths will directly enter the single-arm observational cohort);
4. Subjects or their legally authorized representatives can understand the purpose of the trial, voluntarily participate in the trial and sign informed consent form, and be able and willing to comply with follow-ups and related procedures.

Exclusion Criteria:

1. Subjects with femoral artery occlusion or visually estimated lumen diameter <5mm;
2. Subjects with prior surgical procedures, percutaneous transluminal angioplasty (PTA), stent placement, or vascular grafts at the access site;
3. Subjects with visible calcification at the access site, clinically significant peripheral vascular disease (requiring intervention), or stent implantation ≤1cm from the puncture site;
4. Subjects whose puncture site is above the lowest edge of the inferior epigastric artery and/or above the inguinal ligament as identified by skeletal markers;
5. Subjects with posterior wall vascular puncture or multiple femoral artery punctures due to difficulty in obtaining vascular access;
6. Patients with pathological obesity (BMI >40 kg/m²);
7. Subjects with pre-existing access site complications (hematoma, pseudoaneurysm, arteriovenous fistula, dissection, etc) or any procedure-related complications that may affect recovery, ambulation, or discharge timing;
8. Subjects with acute ST-segment elevation myocardial infarction within 48 hours prior to the procedure;
9. Subjects with uncontrolled hypertension during closure (Systolic BP >180 mmHg or Diastolic BP >110 mmHg);
10. Subjects who are known to be contraindicated or allergic to iodine-containing contrast agents or polyethylene glycol materials;
11. Subjects with severe thrombocytopenia (Platelet count <30×10⁹/L), hemophilia, von Willebrand disease, or severe anemia (Hemoglobin <10 g/dL, Hematocrit <30%);
12. International normalized ratio (INR) >1.5;
13. Subjects with systemic infection or skin infection at the puncture site, or planned indwelling sheath;
14. Subjects unable to ambulate 6 meters without assistance;
15. Pregnant or lactating women;
16. Subjects currently participating in other drug/device clinical trials;
17. Other subjects deemed ineligible for this clinical trial by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Device Success Rate | Intra-procedure

SECONDARY OUTCOMES:
Time to Hemostasis | Time from completion of femoral artery puncture site closure operation using the vascular closure device system to achievement of hemostasis, which will be assessed up to 1 day
Time to Ambulation | Time from completion of femoral artery puncture site closure operation using the vascular closure device system to the patient's ability to ambulate at least 6 meters, which will be assessed up to 30 days
Time to Hospital Discharge | Time from completion of femoral artery puncture site closure operation using the vascular closure device system to Hospital discharge determined by physician, which will be assessed up to 30 days

OTHER OUTCOMES:
Incidence of Major Femoral Access Site Complications within 30 Days Post-Procedure | Up to 37 days
Incidence of Minor Femoral Access Site Complications within 30 Days Post-Procedure | Up to 37 days
Incidence of Device Deficiency | Day 1
Incidence of Adverse Events | Through study completion, an average of 2 months
Incidence of Serious Adverse Events | Through study completion, an average of 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Army Medical University (PLA), Chongqing, China

IPD SHARING:
Plan to Share IPD: No